CLINICAL TRIAL: NCT00451061
Title: The Efficacy of Alpha-blockers for Expulsion of Distal Ureteral Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor449907ctil
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2007-02

CONDITIONS: Renal Colic
Keywords: distal ureterolithiasis; α adrenoreceptors antagonist
MeSH Terms: conditions — Renal Colic | interventions — alfuzosin; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin
Drug: Tamsulosin

SUMMARY:
Most of the patients suffering from renal colic have a distal ureterolithiasis. It had been demonstrated that α adrenoreceptors antagonists, given to patients suffering from renal colic, due to distal ureterolithiasis, had increased the frequency of stone expulsion rate , reduced the time to expulsion and reduced analgesics consumption.Most of the studies evaluated the efficacy of Tamsulosin, which is a selective α 1A and α 1D adrenoreceptors antagonist.(The lower intramural portion of the ureter, where it passes through the detrusor muscle contains mostly α 1D and α 1A adrenergic receptors)

Only one study these days describes the use of Alfuzosin, which is an α adrenergic receptor blocker and not selective for any α 1 adrenergic receptor, for expulsion of distal ureteric stones.Alfuzosin is a drug with a proven efficacy and considered uroselective with high specificity and sensitivity, for the treatment of BPH. There was no significant difference in efficacy between the two α blockers (Alfuzosin vs. Tamsulosin) concerning symptoms relief or flow improvement.

The objective of this study is to compare patient who would receive the standard treatment for distal ureterolithiasis (analgesics, Rowatinex) to patients who would receive also a non selective α blocker (Alfuzosin) or a selective α blocker (Tamsulosin). This in order to evaluate the efficacy of treatment with α blockers for expulsion of distal ureterolithiasis.

DETAILED DESCRIPTION:
The efficacy of alpha-blockers for expulsion of distal ureteral stones

Urolithiasis is estimated among 8%-15% of the population in Europe and North America.1-5 Patient who suffer from renal colic represent a very common reason for visiting the emergency room or for hospitalization. The stones are usually located in the ureter, mostly in its lower third.

Some of the distal ureteral stone would pass spontaneously, depending on a few factors such as the stone's size, location, shape, smooth muscle spasm, submucosal edema and anatomy.

Since renal colic is one of the most painful conditions, the time until expulsion of the stone should be reduced as much as possible. In case the stone obstructs and does'nt pass, damage to the kidney might occur, and surgical intervention should be considered. However, surgery and anesthesia are not risk free.

The local reaction to obstructing ureterolithiasis manifests in ureteric smooth muscle contraction, edema, inflammation and pain. The ureter contains α -adrenergic receptors in the smooth muscle layer, along it's entire length. Since these receptors play an important role in ureteric contraction during renal colic, several studies were performed in order to evaluate the effect of α receptors blockade. These studies had demonstrated that different α blockers had increased the frequency of stone expulsion rate among patients with renal colic, reduced the time to expulsion and reduced analgesics consumption.

Most of the studies evaluated the efficacy of Tamsulosin, which is a selective α 1A and α 1D adrenoreceptors antagonist. The lower intramural portion of the ureter, where it passes through the detrusor muscle contains mostly α 1D and α 1A adrenergic receptors.

A common treatment these days to obstructive uropathy due to benign prostatic hypertrophy (BPH) is Alfuzosin. Despite the fact that it is an α adrenergic receptor blocker and not selective for any α 1 adrenergic receptor subtypes, it is a drug with a proven efficacy and considered uroselective with high specificity and sensitivity, for the treatment of BPH. There was no significant difference in efficacy between the two α blockers (Alfuzosin vs. Tamsulosin) concerning symptoms relief or flow improvement, and side effects were similar.

Only one study these days describes the use of Alfuzosin for expulsion of distal ureteric stones.

The objective of this study is to compare patient who would receive the standard treatment for distal ureterolithiasis (analgesics, Rowatinex) to patients who would receive also a non selective α blocker (Alfuzosin) or a selective α blocker (Tamsulosin). This in order to evaluate the efficacy of treatment with α blockers for expulsion of distal ureterolithiasis.

Materials and methods:

Participants - Individuals who will be referred to the emergency room or be admitted to the urology department in Soroka hospital, (Beer-Sheva, Israel) because of acute renal colic. The patient would be considered for the study only if the stone would be located in the distal ureter.

This study is estimated to include 120 patients and last 6 months. The patients would be divided randomly to three groups:

A. Patients with renal colic that would receive Abitren and Rowatinex B. Same therapy plus Tamsulosin (0.4 mg/daily) C. Same therapy as A plus Alfuzosin (10 mg/daily)

The treatment would last up to 4 weeks.

The duration of the trial would be until expulsion of the stone, but not longer than 4 weeks. Patients who would not pass the stone spontaneously, would be referred to intervention (ESWL, ureteric stent insertion, ureteroscopy)

Treatment discontinuation would be due to hospitalization (intractable pain, fever, the need for an intervention)

The α blockers treatment would be once daily, until stone expulsion, or up to four weeks.

The initial treatment protocol would be the standard treatment - I.V fluids and analgesics

Each patient would be initially evaluated by:

* physical examination
* abdominal radiography
* serum creatinine and leukocytes measurement
* urinalysis
* renal ultrasonography
* blood pressure measurement

The follow up:

The blood pressure measurements would be taken by the family physician, two days and one week after the beginning of the treatment. Four weeks after the treatment begins, each patient would be checked in the out patient clinic. Unenhanced CT scan, serum creatinine and blood pressure measurement would be taken. In case the patient would not pass the stone, intervention would be scheduled.

ELIGIBILITY:
Inclusion Criteria:

• renal colic due to radiologically proven distal ureteral stones

Exclusion Criteria:

* stone larger than 10 mm
* fever
* urinary tract infection
* additional stones, that might be the reason for the renal colic
* severe hydronephrosis
* known sensitivity to α blockers
* concomitant treatment with α blockers, β blockers, calcium antagonists, and nitrates
* pregnancy
* inability to provide informed consent
* a history of surgery or endoscopic procedures in the urinary tract
* history of spontaneous stone expulsion
* known ureteral stricture
* diabetes
* blood pressure values lower than 100/70 mm hg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
frequency of stone expulsion
time to stone expulsion
analgesics consumption

CONTACTS AND LOCATIONS:
Overall Officials: Eran Rosenberg, M.D, Principal Investigator — Soroka university medical center, Beer-Sheva, Israel; Igor Romanowski, M.D, Study Director — Soroka university medical center, Beer-Sheva, Israel
Locations (1):
- Urology department, Soroka university medical center, Beer-Sheva, P,o,box 151, Israel

REFERENCES:
- [Background] De Sio M, Autorino R, Di Lorenzo G, Damiano R, Giordano D, Cosentino L, Pane U, Di Giacomo F, Mordente S, D'Armiento M. Medical expulsive treatment of distal-ureteral stones using tamsulosin: a single-center experience. J Endourol. 2006 Jan;20(1):12-6. doi: 10.1089/end.2006.20.12. PMID 16426124
- [Background] Dellabella M, Milanese G, Muzzonigro G. Randomized trial of the efficacy of tamsulosin, nifedipine and phloroglucinol in medical expulsive therapy for distal ureteral calculi. J Urol. 2005 Jul;174(1):167-72. doi: 10.1097/01.ju.0000161600.54732.86. PMID 15947613
- [Background] Yilmaz E, Batislam E, Basar MM, Tuglu D, Ferhat M, Basar H. The comparison and efficacy of 3 different alpha1-adrenergic blockers for distal ureteral stones. J Urol. 2005 Jun;173(6):2010-2. doi: 10.1097/01.ju.0000158453.60029.0a. PMID 15879806
- [Background] Dellabella M, Milanese G, Muzzonigro G. Efficacy of tamsulosin in the medical management of juxtavesical ureteral stones. J Urol. 2003 Dec;170(6 Pt 1):2202-5. doi: 10.1097/01.ju.0000096050.22281.a7. PMID 14634379
- [Background] Autorino R, De Sio M, Damiano R, Di Lorenzo G, Perdona S, Russo A, Quarto G, Cosentino L, D'Armiento M. The use of tamsulosin in the medical treatment of ureteral calculi: where do we stand? Urol Res. 2005 Dec;33(6):460-4. doi: 10.1007/s00240-005-0508-0. Epub 2005 Nov 29. PMID 16317534
- [Background] Pricop C, Novac C, Negru D, Ilie C, Pricop A, Tanase V. [Can selective alpha-blockers help the spontaneous passage of the stones located in the uretero-bladder junction?]. Rev Med Chir Soc Med Nat Iasi. 2004 Jan-Mar;108(1):128-33. Romanian. PMID 15688769
- [Background] Saita A, Bonaccorsi A, Marchese F, Condorelli SV, Motta M. Our experience with nifedipine and prednisolone as expulsive therapy for ureteral stones. Urol Int. 2004;72 Suppl 1:43-5. doi: 10.1159/000076591. PMID 15133333
- [Background] Micali S, Grande M, Sighinolfi MC, De Carne C, De Stefani S, Bianchi G. Medical therapy of urolithiasis. J Endourol. 2006 Nov;20(11):841-7. doi: 10.1089/end.2006.20.841. PMID 17144848
- [Background] Porpiglia F, Vaccino D, Billia M, Renard J, Cracco C, Ghignone G, Scoffone C, Terrone C, Scarpa RM. Corticosteroids and tamsulosin in the medical expulsive therapy for symptomatic distal ureter stones: single drug or association? Eur Urol. 2006 Aug;50(2):339-44. doi: 10.1016/j.eururo.2006.02.023. Epub 2006 Mar 3. PMID 16574310
- [Background] Beach MA, Mauro LS. Pharmacologic expulsive treatment of ureteral calculi. Ann Pharmacother. 2006 Jul-Aug;40(7-8):1361-8. doi: 10.1345/aph.1G586. Epub 2006 Jul 18. PMID 16849614
- [Background] Lipkin M, Shah O. The use of alpha-blockers for the treatment of nephrolithiasis. Rev Urol. 2006;8 Suppl 4(Suppl 4):S35-42. PMID 17216000
- [Background] Porena M, Guiggi P, Balestra A, Micheli C. Pain killers and antibacterial therapy for kidney colic and stones. Urol Int. 2004;72 Suppl 1:34-9. doi: 10.1159/000076589. PMID 15133331
- See also: Guidelines on benign prostatic hyperplasia,2004,p.36 — http://www.berlin.uroweb.org/